CLINICAL TRIAL: NCT04052581
Title: Assessment of Safety and Outcomes in Patients Undergoing a Standard-of-care Combined POEM-TIF Procedure
Brief Title: Prospective Collection of Outcome Data Post POEM-TIF Procedure
Status: Withdrawn | Type: Observational
Why Stopped: The study is not relevant anymore.
Sponsor: Johns Hopkins University (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00220604
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Achalasia; Gastroesophageal Reflux Disease
Keywords: Per oral Endoscopic Myotomy; Transoral Incisionless Fundoplication; POEM; TIF
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POEM-TIF: All participants will undergo the POEM-TIF in the same session.
  Interventions: Procedure: POEM-TIF

INTERVENTIONS:
Procedure: POEM-TIF — Transoral Incisionless Fundoplication (TIF) following Per oral Endoscopic Myotomy (POEM) in the same session

SUMMARY:
Per Oral Endoscopic Myotomy has been established as a safe and effective treatment of Achalasia type I and II; however, it is limited by post-procedure gastroesophageal reflux. Transoral Incisionless Fundoplication (TIF) has been introduced as the endoscopic gold standard for anti-reflux procedure. Recently, combined POEM-TIF has been performed successfully as a standard of care treatment for patients with severe GER after POEM. We aim to study the safety and feasibility of performing POEM-TIF (POEM and TIF in the same endoscopic session). This study will also put the groundwork for a randomized clinical trial to further study the clinical outcome of the POEM-TIF procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age greater than 18 years old
* Manometrically proven diagnosis of either type I or type II achalasia.

Exclusion Criteria:

* Achalasia type III, or other esophageal dysmotility disorders.
* Completion of POEM with evidence of mucosal injury or compromise
* Previous surgery of the stomach such as sleeve gastrectomy, gastric bypass, Heller myotomy, partial or complete fundoplication, or partial/complete gastrectomy
* Esophageal lumen diameter greater than 4 cm
* Sigmoidization of the esophagus
* Large esophageal diverticula
* Known active gastroesophageal malignancy
* Inability to tolerate sedated upper endoscopy due to cardiopulmonary instability, severe pulmonary disease or other contraindication to endoscopy
* Cirrhosis with portal hypertension, varices, and/or ascites
* Pregnant or breastfeeding women (all women of child-bearing age will undergo urine pregnancy testing)
* Acute gastrointestinal bleeding
* Uncorrectable coagulopathy defined by international normalized ratio (INR) > 1.5 or platelet < 50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient age > 18 years old who have been diagnosis with either type I or type II Achalasia that has been proved by manometry
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Safety of POEM-TIF as assessed by the American Society of Gastrointestinal Endoscopy (ASGE) lexicon scoring system | 6 months
  Safety will be evaluated by the frequency of severe adverse events with probable or definite attribution to the procedure based the ASGE lexicon scoring system. ASGE lexicon's severity grading system classify the adverse events into one of the four categories of mild, moderate, severe, and fatal. Mild adverse event means an adverse event that result in (1) Procedure aborted (or not started) because of an adverse event, (2) Post-procedure medical consultation, or (3) Unplanned hospital admission or prolongation of hospital stay for lesser or equal to 3 nights. Fatal grade adverse event happens when the procedure cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No